CLINICAL TRIAL: NCT01571895
Title: A Phase 2, Multicentre, Single Arm, Pilot Study to Assess the Efficacy and the Safety of 150 mg Twice a Day Oral DF2156A in Patients With Active Bullous Pemphigoid.
Brief Title: Pilot Efficacy and Safety Study of Oral DF2156A in Patients With Active Bullous Pemphigoid
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy observed at 1/3 of the enrollment at investigated dosage. No results available.
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEX0111; 2011-000756-42 (EudraCT Number)
Record Dates: First submitted 2012-04-04; First posted 2012-04-05 (Estimated); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Bullous Pemphigoid
Keywords: Autoimmune inflammatory blistering disorder
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — 2'-((4'-trifluoromethanesulfonyloxy)phenyl)-N-methanesulfonylpropionamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DF2156A 150 mg (Experimental): 150 mg capsule twice a day (every 12 h) for a maximum of 14 days
  Interventions: Drug: DF2156A

INTERVENTIONS:
Drug: DF2156A — DF2156A is a novel small molecule that inhibits the biological activity of the CXC ligand 8 [CXCL8; formerly interleukin (IL)-8] through inhibition of the activation of CXCL8 receptors: CXCR1 and CXCR2. This specific inhibitor stems from a program of drug design of molecules intended to modulate chemokine action.

SUMMARY:
The objective of this clinical trial was to evaluate whether DF2156A has a potential in improving the clinical outcome in patients with active blistering bullous pemphigoid (BP) to warrant its further development. The safety of DF2156A in the specific clinical setting was also evaluated.

DETAILED DESCRIPTION:
The study was a phase 2, multicentre, single arm, pilot study. It has been designed to determine if DF2156A has sufficient activity to warrant its further development.

A total of twelve (12) BP patients were planned to be involved. They were planned to receive DF2156A orally at the dose of 150 mg twice a day for a maximum of 14 days.

Recruitment was intended to be competitive among the study sites, until the planned number of patients is enrolled. Competitive recruitment has been chosen to increase the speed of recruitment and to account for any unexpected occurrence at a site that negatively impact enrolment rate.

The single arm design has been chosen as an appropriate tool for this pilot phase 2 study, considering that BP is a rare disease where a placebo control is not acceptable. Moreover, as there is no spontaneous acute recovery from the active blistering condition, any improvement in patient outcome can be attributed to a positive effect of the Investigational Product.

Each patient was intended to be involved in the study for a screening period, for 14 days of treatment, for all required measurements up to hospital discharge (planned on day 8+1 of treatment) and for one assessment occasion on day 15+1, either during hospital stay or after hospital discharge (out-patient visit). An optional post-treatment visit might be scheduled at day 30+3.

Due to the lack of efficacy observed at 1/3 of the enrollment at the investigated dosage, the patients' enrollment was interrupted and trial, hence, was early terminated. More precisely, only 1 of the 4 enrolled patients completed the study's 14-day treatment period. The remaining 3 patients were discontinued from the study early (1 patient due to treatment failure and 2 patients who were discontinued and admitted to rescue therapy).

While DF2156A appeared to be safe and was generally well-tolerated with only mild AEs reported in 3 patients (and no deaths, SAEs, or discontinuations from the study due to AEs), the limited sample size of the safety population prevents any overall conclusions of safety regarding the investigational product. For this reason no results other than listings are available.

See the MEX0111 synopsis on the EU Clinical Trial Register: https://www.clinicaltrialsregister.eu/ctr-search/rest/download/result/attachment/2011-000756-42/1/27931

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged >50 years.
* Patients with newly diagnosed or relapsing bullous pemphigoid based on clinical diagnosis to be confirmed by direct immunofluorescence and indirect immunofluorescence on salt-spit skin (or BP180 and/or BP230 ELISA). Confirmation by laboratory tests will be obtained ideally before or anyway within one week after enrolment.

For the purpose of this study, clinical relapses are defined as re-appearance of clinical symptoms after the patient had attained remission lasting for more than 3 months without immunosuppressive treatment. In patients with relapsing BP, clinical diagnosis will be confirmed by indirect immunofluorescence or BP180 and/or BP230 ELISA only.

* Patients with mild to moderate active blistering disease (total number of blisters between 1 and 30) whether associated or not with urticarial/eczematous lesions.
* Patients with modified ABSIS score ≤50
* Patients free from any systemic treatments that may affect the course of the disease with the following off-period prior to enrolment:

  1. 3 weeks: steroids, dapsone, tetracyclines, nicotinamide,
  2. 3 months: azathioprine, mycofenolate mofetil, cyclophosphamide, methotrexate, intravenous immunoglobulins, immunoadsorption, TNF antagonists
  3. 12 months: rituximab, leflunomide
* Patients free from any topical treatments other than topical antibiotics and antiseptics in the 4 days prior to enrolment.
* Patients able to comply with the protocol procedures for the duration of the study, including scheduled follow-up visits and examinations.
* Patients able to provide informed consent.

Exclusion Criteria:

* Patients with a Karnofsky rating score <40%.
* Patients with mucosal involvement.
* Patients with moderate to severe renal impairment as per calculated creatinine clearance (CLcr) < 50 mL/min according to the Cockcroft-Gault formula (Cockcroft-Gault , 1976).
* Patients with hepatic dysfunction defined by increased ALT/AST > 3 x upper limit of normal (ULN) and increased total bilirubin > 3 mg/dL [>51.3 μmol/L].
* Patients with hypoalbuminemia defined as serum albumin < 3 g/dL.
* Patients with a baseline (day 0/1, pre-dose) QTcF > 470 msec.
* Patients who had a myocardial infarction in the 6 months prior to enrolment.
* Patients on treatment with phenytoin, warfarin, sulphonylurea hypoglycemics (e.g. tolbutamide, glipizide, glibenclamide/glyburide, glimepiride, nateglinide) and high dose of amitriptyline (> 50 mg/day).
* Patients with known hypersensitivity to non-steroidal antiinflammatory drugs.
* Patients using any investigational agent within 12 months prior to enrolment.
* Pregnant or breast feeding women. Unwillingness to use effective contraceptive measures up to 2 months after the end of study drug administration (females and males).

Additional Exclusion Criteria for Germany only:

* Patients with hypokalemia defined as serum potassium < 3.5 mmol/L.
* Patients with clinically relevant bradycardia (heart rate < 50 beats/min)
* Patients with a complete left bundle branch block.
* Patients with a history of uncontrolled or labile hypertension
* Patients with a history of congestive heart failure.
* Patients with a history of cardiomyopathy.
* Patients with unstable angina pectoris.
* Patients with a personal or family history of congenital or documented acquired QT interval prolongation.
* Patients with a significant atrial or ventricular arrhythmia or symptomatic arrhythmia in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-02-20 (Actual); Primary Completion 2012-07-05 (Actual); Study Completion 2012-07-05 (Actual)

PRIMARY OUTCOMES:
Total number of blisters from baseline | day 0/1 (pre-dose), 8 and 15
  Total number of blisters from baseline
Modified ABSIS score change from baseline | day 0/1 (pre-dose), 8 and 15
  ABSIS score will be measured according to the pemphigus scoring sheet [Rosenbach, 2009] adjusted to the clinical manifestation in BP patients, as per specifications in protocol.
Physician Global Assessment (PGA) score measured on a 0-10 scale [Rosenbach, 2009]. Percent change from baseline | day 0/1 (pre-dose), 8 and 15
  PGA score will be measured according to the following scale:
  0
  1 2 3 4 5 6 7 8 9 10 Perfect Worst health skin condition imaginable
  The following guidelines will help standardize PGA:
  0: no lesions 2: almost cleared, no functional impairment 4: few lesions / low functional impairment 6: moderate 8: severe / extensive 10: life-threatening
Pruritus measured on a 10 cm visual analogue scale. Absolute value change from baseline | day 0/1 (pre-dose), 8 and 15
  Pruritus will be measured according to the following scale:
  0 10 No pruritus Worst pruritus I can imagine
Eosinophil blood count. Percent change from baseline | screening and day 15
  Eosinophil blood count. Percent change from baseline
Percentage of patients with treatment failure (drug discontinuation due to disease worsening) | day 8
  treatment failure (drug discontinuation due to disease worsening)
Percentage of patients completely free from blisters | day 15
  Percentage of patients completely free from blisters
Number of patients who are still free from blisters without requiring any systemic or topical rescue treatment - Optional | Day 30
  Number of patients who are still free from blisters without requiring any systemic or topical rescue treatment - Optional
QTcF. Change from baseline | Italy: day 0/1 (pre-dose), day 1, 5, 8 and 15___Ger:day 0/1 (pre-dose), day 1, 3, 5, 8 and 15
  QTcF. Change from baseline
Incidence of Adverse Events and Serious Adverse Events | throughout the study up to day 15 or 30
  Incidence of Adverse Events and Serious Adverse Events
Blisters percent change from baseline | day 0/1 (pre-dose), 8 and 15
  Blisters percent change from baseline
Modified ABSIS score percent change from baseline | day 0/1 (pre-dose), 8 and 15
  ABSIS score will be measured according to the pemphigus scoring sheet [Rosenbach, 2009] adjusted to the clinical manifestation in BP patients, as per specifications in protocol.
Physician Global Assessment (PGA) score measured on a 0-10 scale [Rosenbach, 2009]. Absolute value change from baseline | day 0/1 (pre-dose), 8 and 15
  PGA score will be measured according to the following scale:
  0
  1 2 3 4 5 6 7 8 9 10 Perfect Worst health skin condition imaginable
  The following guidelines will help standardize PGA:
  0: no lesions 2: almost cleared, no functional impairment 4: few lesions / low functional impairment 6: moderate 8: severe / extensive 10: life-threatening
Pruritus measured on a 10 cm visual analogue scale. Percent change from baseline | day 0/1 (pre-dose), 8 and 15
  Pruritus will be measured according to the following scale:
  0 10 No pruritus Worst pruritus I can imagine
Eosinophil blood count. Absolute number change from baseline | screening and day 15
  Eosinophil blood count. Absolute number change from baseline
Number of patients with treatment failure (drug discontinuation due to disease worsening) | day 8
  Number of patients with treatment failure (drug discontinuation due to diseas
Number of patients completely free from blisters | day 15
  Number of patients completely free from blisters
QTcF. Absolute value | Italy: day 0/1 (pre-dose), day 1, 5, 8 and 15___Ger:day 0/1 (pre-dose), day 1, 3, 5, 8 and 15
  QTcF. Absolute value

SECONDARY OUTCOMES:
Plasma levels of DF2156A and its major metabolites (DF2227 and DF2108) at steady state conditions | day 5 and 8
  Plasma levels of DF2156A and its major metabolites (DF2227 and DF2108) at steady state conditions

CONTACTS AND LOCATIONS:
Overall Officials: Biagio Didona, MD, Principal Investigator — I Divisione di Dermatologia, Istituto Dermopatico dell'Immacolata, IRCCS; 00167 Roma, Italy; Detlef Zillikens, MD, Principal Investigator — Klinik für Dermatologie, Allergologie und Venerologie - Univ. Schleswig-Holstein; Lübeck, Germany; Andrea Kneisel, MD, Principal Investigator — Klinik für Dermatologie und Allergologie - Philips Universität; 35037 Marburg, Germany; Johannes Kern, MD, Principal Investigator — Department of Dermatology - Universitäts-Hautklinik; 79104 Freiburg, Germany; Pier Adelchi Ruffini, MD, Study Director — Development Director Dompé s.p.a., 20122 Milan, Italy
Locations (4):
- Germany (3):
  - Department of Dermatology - Universitäts-Hautklinik; Hauptstraße 7, Freiburg im Breisgau
  - Klinik für Dermatologie, Allergologie und Venerologie - Universitätsklinikum Schleswig-Holstein, Campus Lübeck; Ratzeburger Allee 160, Lübeck
  - Klinik für Dermatologie und Allergologie - Philips Universität; 35037, Marburg
- I Divisione di Dermatologia, Istituto Dermopatico dell'Immacolata, IRCCS;, Roma, Italy